CLINICAL TRIAL: NCT06781983
Title: A Phase 1, Open-label, Multi-center Study of the Safety, Tolerability, and Efficacy of IPH4502 as a Single Agent in Advanced Solid Tumors
Brief Title: Safety and Tolerability of IPH4502 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH4502-101
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Exatecan; Topo-Isomerase I inhibitor; Squamous cell carcinoma of the head and neck; Esophageal squamous cell carcinoma; Triple negative breast cancer; Non-small cell lung cancer; Gastro-esophageal junction and gastric cancer; Colorectal carcinoma; Ovarian carcinoma; Prostate cancer; Cervical cancer; Melanoma; Urothelial carcinoma; Antibody-drug conjugates; ADC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Uterine Cervical Neoplasms; Melanoma; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IPH4502 Monotherapy (Experimental)
  Interventions: Drug: IPH4502

INTERVENTIONS:
Drug: IPH4502 — Part 1 (dose escalation) and Part 2 (dose optimization)

SUMMARY:
This is a first-in-human, open-label, multicenter, Phase 1 study to evaluate the safety, tolerability and preliminary efficacy of IPH4502 and to determine the recommended Phase 2 dose (RP2D) in advanced solid tumors that are known to express Nectin-4

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multicenter, single-arm Phase 1 study, with a part 1 dose escalation guided by a Bayesian optimal interval design with backfilling (BOIN-BF), followed by a part 2 dose optimization in up to 2 selected indications. This study is to measure the safety, tolerability, pharmacokinetics, and preliminary efficacy of escalating doses of IPH4502 in patients with advanced solid tumors that are known to express Nectin-4.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed, unresectable, locally advanced or metastatic solid tumors that are known to express Nectin-4
* Prior systemic treatment for locally advanced or metastatic disease, yet no therapy with demonstrated clinical benefit for the tumor type is available.
* Measurable disease according to RECIST 1.1.
* Archival tumor tissue obtained within 4 months of screening and since the last anticancer therapy prior to the study or agree to undergo a tumor biopsy at baseline.
* Adequate organ function and hematological function.

Main Exclusion Criteria:

* Known or suspected brain metastases.
* Participants with an active infection, Any other infection requiring systemic treatment or latent infection.
* Participants with clinically significant comorbidity(s).
* History of treatment for, or suspicion or confirmed interstitial lung disease (ILD) at baseline.
* Condition being treated with systemic corticosteroids or immunosuppressive therapy during IPH4502 treatment.
* Thromboembolic event requiring anticoagulation therapy ≤14 days prior to the first dose of IPH4502.
* Clinically significant cardiovascular disease and/or cardiac repolarization abnormality.
* Participants with symptomatic heart failure, Acute coronary syndromes
* Participant is receiving or has received anticancer therapy prior to enrolment that may have impact on the assessment of IPH4502.
* Major surgery ≤28 days and minor surgery ≤7 days prior to first dose of IPH4502 or 6 months for coronary artery bypass surgery.
* Concomitant medications or vaccines : Live-attenuated vaccines ≤ 6 weeks prior to first dose of IPH4502; systemic corticosteroids or other immunosuppressive agents within 14 days prior to the first dose of IPH4502; systemic use of moderate or strong CYP 3A4 inhibitors; systemic use of moderate or strong CYP 3A4 inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | From time of first dose through treatment period, including the follow-up: up to 24 months
  To evaluate the incidence of AEs, SAEs, TEAEs, and DLTs.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | From time of informed consent through treatment period, including the follow-up: up to 24 months
  To characterize and evaluate the pharmacokinetic profile of IPH4502.
Area Under the Plasma Concentration (AUC) | From time of informed consent through treatment period, including the follow-up: up to 24 months
  To characterize and evaluate the pharmacokinetic profile of IPH4502.
Incidence of antidrug antibodies (ADA) against IPH4502 | From time of informed consent through treatment period, including the follow-up: up to 24 months
  To evaluate the immunogenicity of IPH4502.
Objective Response Rate (ORR) | From time of informed consent through treatment period, including the follow-up: up to 24 months
  To investigate any preliminary antitumor activity of IPH4502.
Duration Of Response (DoR) | From time of informed consent through treatment period, including the follow-up: up to 24 months
  To investigate any preliminary antitumor activity of IPH4502.
Progression Free Survival (PFS) | From time of informed consent through treatment period, including the follow-up: up to 24 months
  To investigate any preliminary antitumor activity of IPH4502.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Massachusetts General Hospital - Boston, Boston, Massachusetts
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Mount Sinai Tisch Cancer Center, New York, New York
  - NEXT Oncology - Dallas, Dallas, Texas
  - NEXT Oncology - Virginia, Fairfax, Virginia
- France (2):
  - Centre Léon Bérard, Lyon
  - Gustave Roussy Cancer Institute, Villejuif

IPD SHARING:
Plan to Share IPD: No